CLINICAL TRIAL: NCT04575883
Title: High Intensity Interval Training in Youth With Congenital Heart Disease: A Prospective Clinical Trial of a Novel Telemedicine Video Game-Linked Exercise Platform
Brief Title: HIIT in Youth With Congenital Heart Disease (MedBIKE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00102421
Record Dates: First submitted 2020-08-28; First posted 2020-10-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Congenital Heart Disease; Pediatric ALL
Keywords: Cardiac rehabilitation; High Intensity Interval Training; Telemedicine
MeSH Terms: conditions — Heart Defects, Congenital; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MedBIKE HIIT (Experimental): MedBIKE HIIT Exercise Program
  Interventions: Device: MedBIKE HIIT

INTERVENTIONS:
Device: MedBIKE HIIT — Participants will complete a high intensity interval training exercise program 3 times a week for 12 weeks (36 sessions total)

SUMMARY:
Congenital heart disease (CHD), the most common birth defect, is present in nearly 1% of the population. CHD patients are associated with intense resource utilization and premature death in adulthood. The risk of premature death is linked with reduced exercise capacity, a finding consistently noted in youth with CHD. Reduced exercise capacity in this population has also been associated with reduce physical activity and health-related quality of life.

Cardiac rehabilitation (CR) in adults with acquired heart disease is an established secondary prevention strategy that improves exercise capacity. The investigators propose a prospective clinical trial of a home-based high intensity interval training (HIIT) program using a novel telemedicine-equipped video game-linked cycle ergometer (MedBIKE™) for 10 to 18 year olds with repaired moderate-complex CHD. The pilot study with the MedBIKE has shown promising results. The investigators now seek to study the efficacy of this program in a broader CHD population.

DETAILED DESCRIPTION:
Purpose: This project is a prospective clinical trial of a home-based high intensity interval training (HIIT) exercise program using a novel telemedicine-enabled and video game-linked customizable cycle ergometer (MedBIKE™) in the pediatric congenital heart disease (CHD) population.

Hypothesis: The home-based the MedBIKE™ HIIT program will significantly improve exercise capacity. The MedBIKE intervention will significantly improve time spent in MVPA and reduce sedentary time, improve HRQoL and self-efficacy towards PA, and improve endothelial function. Moreover, the investigators hypothesize that the improvements in exercise capacity, along with the improvements in the secondary outcomes will remain significantly improved up to one-year post- MedBIKE intervention, when compared to pre-intervention values.

Justification: Exercise intervention studies in the pediatric CHD population have been limited by small sample sizes and there is limited data pertaining to the sustained effects of exercise interventions on exercise capacity, physical activity, endothelial function, and quality of life. This study, using standardized and largely operator-independent measure, will be one of the largest exercise intervention clinical trials in the pediatric CHD population.

Primary Objective: Evaluate the impact of an eight-week, home-based HIIT MedBIKE™ program on exercise capacity in youth with repaired moderate-complex CHD.

Secondary Objectives: Evaluate the impact of the MedBIKE™ intervention on 1) PA; 2) HRQoL and self-efficacy towards PA; 3) endothelial function; and 4) sustained changes in the primary and secondary outcomes.

Research Method: This will be a single-center, prospective clinical trial. Potential participants and families will be approached first by a clinical team member. In addition, flyers with key study information will be placed in waiting rooms of the pediatric cardiology clinics. Participants and parents expressing interest will meet with a research coordinator who, along with one of the investigators and the clinical team will screen for eligibility. Written consent and assent (if applicable) will be obtained from participants who are deemed eligible.

Following recruitment, participants will be administered the TACQOL and CSAPPA questionnaires and an accelerometer to be worn for 7-days, after which participants will arrive for the baseline assessment. As participants must be NPO for EndoPAT testing, they will have a small meal following EndoPAT testing and at least two hours prior to CPET testing. A MedBIKE will be installed in the participants home within 2-weeks of the baseline CPET at which time an orientation session will occur to review the manual, safety procedures and the telemedicine component. Participation will consist of a 12-week, 3-times per week (36 sessions in total) HIIT program. All sessions will be supervised by an exercise physiologist. Protocol completion will be considered a minimum of 27 of the 36 sessions (75%). Following the completion of the intervention, the MedBIKE will be removed by the participants home and returned to the Stollery Children's Hospital.

A follow-up assessment, identical to that of the baseline (questionnaires, EndoPAT, CPET, interviews and a 7-day week wear of an accelerometer) will occur 3-14 days post-intervention. These assessments will be repeated at 6- and 12-months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 10-18 years
* Repaired moderate-complex congenital heart disease

Exclusion Criteria:

* Non-English speaking (thus limiting communication during the MedBIKE™ sessions)
* Home environment cannot accommodate the MedBIKE™ system (space limitations)
* Previous involvement in a cardiac rehab or exercise intervention program
* Primary cardiologist has exercise restricted the participant or counsels against participation
* Previous exercise stress test demonstrating sustained arrhythmias, ST segment elevation or depression greater than 3mm, an inappropriate rise in blood pressure (BP) (<20 mmHg) or a systolic BP >200 mmHg, or symptoms of chest pain or syncope
* Resting arterial saturation <85% or oxygen requirements
* Moderate ventricular systolic dysfunction (or worse) at the most recent echocardiogram
* History of chest pain on exertion
* Unrepaired/unpalliated CHD
* Arrhythmias in the last year (including supraventricular tachycardia, ventricular tachycardia, atrioventricular block (Mobitz II or worse))
* New York Heart Association class II or worse symptoms
* Active medical inter-current illness limiting ability to participate
* Cognitive impairment limiting the communication needed for the HIIT program
* Extracardiac or congenital abnormality limiting the participant's functional ability to exercise

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity in the change in VO2peak (mL/kg/min) measured through CPET testing | Baseline, 1-week post-intervention, 6-months post-intervention, 12-months post-intervention
  CPET (Exercise Stress Test and Spirometry) will be done to measure the VO2peak (mL/kg/min) output of participants. A comparison will be done pre- and post-MedBIKE intervention, as well as 6 and 12-months post, to determine the change in overall VO2peak of participants. We will also evaluate changes in VE/VCO2, peak power output (W), and HRmax (maximum heart rate).

SECONDARY OUTCOMES:
Changes in physical activity, defined as time spent in moderate to vigorous physical activity (MVPA) and sedentary time, measured by wearing an accelerometer for 7-days prior and 7-days post MedBIKE intervention | Baseline, 1-week post-intervention, 6-months post-intervention, 12-months post-intervention
  Participants will be provided with an accelerometer to wear for 7-days prior to the start of the MedBIKE intervention program and again for 7-days post intervention and again at 6 and 12-months post intervention. The accelerometer will measure the time spent in moderate to vigorous physical activity (MVPA) and the sedentary time. A comparison will be done pre- and post-MedBIKE intervention to determine changes in the physical activity levels. The 6-month and 12-month time points will be used for a comparison on the sustained changes of the intervention.
Changes in Health-Related Quality of Life as measured using the TNO AZL Children's Quality of Life (TACQOL) questionnaire. | Baseline, 1-week post-intervention, 6-months post-intervention, 12-months post-intervention
  Participants will be asked to complete the TNO AZL Children's Quality of Life (TACQOL) questionnaire. This questionnaire is a validated multidimensional instrument to assess the health-related quality of life in youth. The overall score of this questionnaire will be compared pre- and post-MedBIKE intervention to determine changes in health-related quality of life. The 6-month and 12-month time points will be used for a comparison on the sustained changes of the intervention.
Changes in self efficacy towards physical activity measured on the Children's Self-Perceptions of Adequacy in and Predilection for Physical Activity (CSAPPA) scale. | Baseline, 1-week post-intervention, 6-months post-intervention, 12-months post-intervention
  Participants will be asked to complete the Children's Self-Perceptions of Adequacy in and Predilection for Physical Activity (CSAPPA) scale. This questionnaire is a validated tool designed to assess self-perceptions of adequacy and predilection towards physical activity in youth. The overall score of this questionnaire will be compared pre- and post-MedBIKE intervention and again at 6 and 12-months post-intervention to evaluate sustained changes.
Changes in endothelial function to determine arterial volume will be measured using an EndoPAT 2000 instrument. | Baseline, 1-week post-intervention, 6-months post-intervention, 12-months post-intervention
  Changes in endothelial function will be measured using an EndoPAT 2000. The EndoPAT is an observer-independent assessment that evaluates changes in arterial volume via finger plethysmography by capturing beat-to-beat variations in arterial pulse wave amplitude, thus generating a peripheral arterial tone (PAT) signal. The EndoPAT score will be compared pre- and post-MedBIKE intervention and again at 6 and 12-months post-intervention to evaluate sustained changes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Khoury, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers. All data will be de-identified prior to analysis and published.

REFERENCES:
- [Background] Khoury M, Phillips DB, Wood PW, Mott WR, Stickland MK, Boulanger P, Rempel GR, Conway J, Mackie AS, Khoo NS. Cardiac rehabilitation in the paediatric Fontan population: development of a home-based high-intensity interval training programme. Cardiol Young. 2020 Oct;30(10):1409-1416. doi: 10.1017/S1047951120002097. Epub 2020 Jul 27. PMID 32716280